CLINICAL TRIAL: NCT05606484
Title: Effect of Virtual Reality Exercise on Hemodialysis Patients: A Randomized Controlled Clinical Trial Research Protocol
Brief Title: Effect of Exercise With Virtual Reality in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: European University of Madrid (Other)
Responsible Party: Principal Investigator, Érika Meléndez Oliva, Principal Investigator, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TFM.MMC.EJPP.EMO.220221
Record Dates: First submitted 2022-09-25; First posted 2022-11-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Kidney Failure, Chronic
Keywords: Kidney Failure, Chronic; Inflammation; Functional capacity; Psychological state; Renal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Experimental, controlled and randomized study, whose methodology complies with the CONSORT standards for clinical trials
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients and the evaluator will be blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG) (Experimental): They will perform an intradialysis physical exercise program with non-immersive virtual reality during the first two hours of hemodialysis treatment (n = 40).
  Interventions: Other: Exercise with non-immersive virtual reality; Other: Exercise with a static pedal
- Control Group (CG) (Active Comparator): They will exercise with a static pedal during the first two hour of hemodialysis treatment (n = 40).
  Interventions: Other: Exercise with non-immersive virtual reality; Other: Exercise with a static pedal

INTERVENTIONS:
Other: Exercise with non-immersive virtual reality — Patients will exercise for 30 minutes with non-immersive virtual reality (VR) with a perceived exertion between 12-15 (somewhat hard-hard) on the Borg scale. Patients will perform 3 weekly sessions during the second hour of hemodialysis, on simultaneous days.
Other: Exercise with a static pedal — Patients will exercise with a stationary pedal for 30 minutes at an intensity of 12-15 (somewhat hard-hard) on the Borg scale of perceived exertion. The patients will carry out an exercise session 3 times a week on alternate days, coinciding with the patients of the exercise with VR.

SUMMARY:
Background. An increase in inflammatory biomarkers is associated with impaired kidney function and increased cardiovascular risk and mortality. Physical exercise has been shown to improve the functional capacity and inflammatory status of patients undergoing hemodialysis (HD) treatment, increasing their health-related quality of life. Virtual reality (VR) is an effective and safe tool to increase patient adherence to the exercise program, however, there are very few studies that analyze its effect on the functional capacity of patients with chronic kidney disease (CKD) in HD and none analyze its effect on the inflammatory state of these patients, which justifies the performance of this study.

Methods. Eighty patients with CKD on HD treatment will be randomly assigned into two groups, one of them will perform an intradialysis exercise program with non-immersive VR (intervention group; n=40), and the other will exercise with a static pedal (control group; n). =40). The functional capacity of the patients and their inflammatory and psychological status, as well as their exercise adherende, will be analyzed before and after exercise programs.

DETAILED DESCRIPTION:
Description of the intervention The exercise program will last for 12 weeks. Randomly, half of the patients will be instructed to - Control Group (CG): They will be instructed to exercise with a static pedal (control group) and the other half will be instructed to carry out the intradialysis non-immersive virtual reality exercise program.

* Intervention Group (IG): Will perform an intradialysis physical exercise program with non-immersive virtual reality during the first two hours of hemodialysis treatment (n = 40).
* Control Group (CG): They will exercise with a static pedal (n = 40). Exercise program The direction and supervision of the exercise programs will be the responsibility of the nursing staff of the Hemodialysis Unit and several physiotherapists of the Rehabilitation Unit of the General University Hospital of Alicante Doctor Balmis, the nursing staff being in charge of directing and supervising the intradialysis exercise program.

Prior to the beginning of the intervention, said personnel will receive exhaustive training on the characteristics of the exercise program and on how to carry it out in an optimal way. In this training they will be instructed on how to execute each of the exercises in the program with virtual reality.

During the two weeks prior to the intervention, a "first contact" period will be carried out, during which the nursing staff will implement the virtual reality intradialis exercise program as a test, so that they can familiarize themselves with the material necessary to exercise, as well as resolve any doubts that may arise. This trial period will be supervised by the physiotherapist in charge of giving them the training.

On the other hand, to improve adherence to exercise by patients and avoid losses throughout the program, all the staff in charge of directing and supervising the exercise will receive a training session by a psychologist specialized in managing barriers in special populations during exercise, with the aim of developing strategies to address these barriers during the intervention period.

The exercise program will have a duration of 12 weeks, with a frequency of 3 exercise sessions per week, these being of a progressive duration according to the patient's capacity (EEP 13-15), until reaching 30 minutes per session, and performed during the first two hours of HD treatment.

Before and after each exercise session, heart rate and blood pressure will be recorded.

Patients will be instructed to perform the exercise independently or with minimal assistance.

The non-immersive virtual reality exercise program is described below:

- Intervention Group (IG): Participants assigned to this group will start with a 5-minute warm-up session and then perform a virtual reality exercise session for up to a maximum of 30 minutes, depending on the rate of perceived exertion that should be felt between "somewhat hard" and "hard" (13-15 out of 20 in EEP). The intensity will progress by increasing the number of exercise series (each lasting 3 minutes) and may vary between 1 and 10 series, depending on the patient's capacity, taking a 1-minute break between each series.

The hemodialysis session may be carried out simultaneously with the exercise, since the work will focus on the lower limbs.

An adapted version of ACT (Treasure Hunt) will be used for the VR program. ACT is a non-immersive virtual reality system designed with a playful scheme. For the participants, the system is an intradialysis virtual reality game, which makes dialysis sessions more enjoyable. In ACT, the subject tries to hit a series of targets (avoiding obstacles) by moving the leg.

The difficulty in ACT is graduated according to the characteristics of the participants, who will be able to change the leg during the game when they feel tired.

The general hardware setup consists of a standard computer, a television (commonly found in HD units), and a Ms Kinect® motion tracking system.

At the beginning of the session, the therapists define the VR intervention for the session using a management tool, adding different rest periods and configuring their duration. The difficulty level of the exercise will also be set at startup, and therapists will be able to program the system to automatically increase or decrease the difficulty level depending on the participant's performance.

Before their first session, each participant will receive instructions on the general use of the system and a test session will take place.

At the end of the program, participants will end the session with another 5 minutes of gentle stretching.

Control group (CG): The participants in this group will exercise with a static pedal, exercising the same muscle groups as the VR group. They will perform the exercise at the same time as the VR group, during the first two hours of hemodialysis, with a duration of 30 minutes each session, performing 3 weekly sessions at a perceived exertion intensity of 12-15 (something hard-hard) in the Borg scale.

The patients will be blind, being distributed in the hemodialysis room so that in one area there are the patients who exercise with VR and in the other the patients who exercise with a static pedal.

ELIGIBILITY:
Inclusion criteria:

- Patients with CKF in a stable clinical situation who have been on HD treatment for at least 3 months.

Exclusion criteria:

* Had a myocardial infarction in the 6 months before the start of the study
* Suffered unstable angina at rest or during exercise
* Have cerebrovascular diseases (such as transient ischemia or stroke)
* Present amputation of lower limbs above the knee without prothesis
* Present a musculoskeletal or respiratory pathology likely to worsen with exercise
* Present an inability to carry out functional assessment tests
* Present visual or cognitive impairments that affect the ability to use the VR equipment or understand the VR exercise

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-09 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of Interleuquine 6 (IL-6) (pg/ml) | Change from Baseline IL-6 at 12 weeks
  Inflammatoy marker
Change of Tumoral Necrosis Factor-alpha (TNF-alpha) (pg/ml) | Change from Baseline TNF-a at 12 weeks
  Inflammatoy marker
Change of C Reactive Protein (CRP) (mg/L) | Change from Baseline CRP at 12 weeks
  Inflammatoy marker
Change of Intercellular Adhesion Molecule 1 (ICAM 1) (ng/ml) | Change from Baseline ICAM 1 at 12 weeks
  Inflammatoy marker
Change of Vascular cell adhesion protein 1 (VCAM 1) (ng/ml) | Change from Baseline VCAM 1 at 12 weeks
  Inflammatoy marker

SECONDARY OUTCOMES:
Assessment of the functional capacity of patients: Short Physical Performance Battery (SPPB) | baseline and up to 12 weeks
  Mesure dependency, institutionalization, hospitalization and mortality. Score ranges from 1 to 12 points
Assessment of the functional capacity of patients: 10 Sit To Stand Test (10 STS). | baseline and up to 12 weeks
  Seconds it takes for the patient to get up and sit down 10 times
Assessment of the functional capacity of patients: 60 Sit To Stand Test (60 STS). | baseline and up to 12 weeks
  Number of times the patient gets up and sits down during 60 seconds
Assessment of the functional capacity of patients: 6 minute walk test (6MWT) | baseline and up to 12 weeks
  Meters that a patient is able to walk for 6 minutes
Psychological assessment of patients: Multidimensional Questionnaire of Adaptation to the Disease for Renal Patients on Dialysis | baseline and up to 12 weeks
  It consists of two phases: Phase A and Phase B. The Phase A, which includes 12 items, collects all the information from the clinical history of the patient. This phase includes two areas "Data Doctors" and "Previous Psychopathological History". Phase B, which includes 51 items, it is made up of nine areas that make up the evaluation of the patient. This phase includes the following areas: "Sociodemographic data" (6 items), "Information",(9 items), "Medication and diet" (3 items), "Social support" (4 items), "State of encouragement" (2 items), "Personal resources, coping and resilience" (8 items), "Learning and perceived changes" (5 items), "Spirituality" (2 items) and "Care planning" (2 items). The questions have four formats of response; three of them closed in nature (dichotomous responses, nominal categorical, and 10-point Likert-type scales), and one open and qualitative. An increase in the scale score is positive. A change α < 0.05 is considered statistically significant.

IPD SHARING:
Plan to Share IPD: No